CLINICAL TRIAL: NCT00005625
Title: Phase II Study of ET-743 Therapy in Metastatic Osteosarcoma
Brief Title: Ecteinascidin 743 in Treating Patients With Previously Treated Metastatic Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-098; CDR0000067769 (Registry Identifier: PDQ (Physician Data Query)); PMAR-ET-019-99; NCI-G00-1761
Record Dates: First submitted 2000-05-02; First posted 2004-04-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Sarcoma
Keywords: metastatic osteosarcoma; recurrent osteosarcoma
MeSH Terms: conditions — Sarcoma; Osteosarcoma | interventions — Trabectedin

INTERVENTIONS:
Drug: trabectedin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of ecteinascidin 743 in treating patients who have previously treated metastatic osteosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the partial and complete response rate in patients with previously treated metastatic osteosarcoma when treated with ecteinascidin 743. II. Further characterize the toxicity profile and the pharmacokinetic-pharmacodynamic relationships of this drug in this patient population.

OUTLINE: This is a multicenter study. Patients receive ecteinascidin 743 IV over 24 hours. Treatment continues every 6 weeks in the absence of unacceptable toxicity or disease progression for at least 2-6 courses. Patients with a complete response (CR) receive at least 2 additional courses after documented CR. Patients are followed every 3 months until disease progression. All patients are followed until death after disease progression.

PROJECTED ACCRUAL: A total of 25-33 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven osteosarcoma previously treated with standard chemotherapy agents (methotrexate, doxorubicin/cisplatin, ifosfamide) Active metastatic disease following chemotherapy At least 1 bidimensionally measurable lesion located in a nonirradiated area CT scan lesion at least 20 mm in at least 1 diameter Clinically measurable lesion at least 20 x 20 mm No symptomatic or known brain or leptomeningeal involvement

PATIENT CHARACTERISTICS: Age: 12 and over Performance status: WHO 0-1 Life expectancy: At least 3 months Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) Alkaline phosphatase no greater than ULN OR Alkaline phosphatase liver fraction and 5'-nucleotidase no greater than ULN AST/ALT less than 2.5 times ULN Albumin greater than 25 g/L No clinically significant liver disease Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 40 mL/min Cardiovascular: No congestive heart failure or angina pectoris even if medically controlled No myocardial infarction within past year No uncontrolled arterial hypertension No arrhythmias Other: Not pregnant or nursing Fertile patients must use effective contraception No history of other malignancy except basal cell carcinoma or carcinoma in situ of the cervix No other serious illness or medical conditions (e.g., history of significant neurological or psychiatric disorders, active infection) No concurrent grapefruit consumption on a regular basis

PRIOR CONCURRENT THERAPY: Biologic therapy: Recovered from prior immunotherapy No concurrent prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF) Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy and recovered No other concurrent local or systemic chemotherapy Endocrine therapy: Not specified Radiotherapy: Recovered from prior radiotherapy No concurrent palliative or primary radiotherapy Surgery: Not specified Other: At least 30 days since other prior investigational drugs No other concurrent investigational drugs No concurrent participation in another clinical trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-12; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gorlick, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States